CLINICAL TRIAL: NCT04626739
Title: An Open, Uncontrolled, Multicenter Clinical Trial to Explore the Safety, Efficacy, and Remission Phase of Chimeric Antigen Receptor T Cell (CAR-T) in the Treatment of Relapsed Refractory (R/R) Non-Hodgkin Lymphoma (NHL)
Brief Title: CAR-T Cells in Treating Patients With Relapsed or Refractory NHL
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T for NHL
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Refractory Indolent Adult Non-Hodgkin Lymphoma
MeSH Terms: interventions — fludarabine; Influenza Vaccines; Cyclophosphamide; Cholestanetriol 26-Monooxygenase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteers (Experimental): The patient voluntarily signs the informed consent, and the patient meets the entry criteria to diagnose patients with Relapsed Refractory (R/R) non-Hodgkin lymphoma
  Interventions: Drug: CD19 CAR-T; Drug: CD22 CAR-T; Drug: CD19+CD22 CAR-T; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CD19 CAR-T — CD19 CAR-T for CD19 positive R/R non-Hodgkin lymphoma
  Other Names: Senl_19
Drug: CD22 CAR-T — CD22 CAR-T for CD22 positive R/R non-Hodgkin lymphoma
  Other Names: Senl_22
Drug: CD19+CD22 CAR-T — CD19+CD22 CAR-T for CD19 positive and CD22 positive R/R non-Hodgkin lymphoma
  Other Names: Senl_19+22
Drug: Fludarabine — 25mg/㎡ for D-4、D-3 and D-2
  Other Names: flu
Drug: Cyclophosphamide — 500mg/㎡ for D-3 and D-2
  Other Names: ctx

SUMMARY:
This is an open, single-arm, phase I clinical study to evaluate efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) in the treatment of Non-hodgkin's lymphoma. A total of 100 patients are planned to be enrolled over a period of 3 years.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells targeted against CD19 have demonstrated unprecedented successes in treating patients with hematopoietic and lymphoid malignancies. In this study, investigators will evaluate their safety and efficacy in patients with different types of hematopoietic and lymphoid malignancies. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, tumor targeting and disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily sign the informed consent, and are willing and able to comply with the visit, treatment protocol, laboratory examination and other requirements of the study as set out in the trial procedure sheet;
2. Cd19-positive R/R NHL patients: recurrent or refractory patients were defined as diffuse large B cell lymphoma (DLBCL), follicular lymphoma (FL), mantle cell lymphoma (MCL), mucosa-associated lymphoid tissue lymphoma (MALTL), and Burkit lymphoma (BL) diagnosed by histopathology.

   To standard treatment for primary drug resistance, or after treatment for at least two line standard specification treatment of PD, or the last treatment effect for SD and duration less than 6 months, or CD20 positive patients by the resistance against CD20 single treatment is invalid or has a relapse, or autologous hematopoietic stem cell transplantation in PD or 12 months after the confirmed by biopsy has a relapse, or to save patients after autologous hematopoietic stem cell transplantation for at the end of the line no ease or relapse after treatment;
3. There should be at least one measurable tumor focal point;
4. Karnofsky [2] score 50 or more;
5. Tumor cells were CD19 positive by immunohistochemistry or flow cytometry;
6. The expected survival time is greater than 3 months;
7. Pregnancy tests for women of childbearing age must be negative; Both men and women should agree to use effective contraceptives during treatment and for the following 1 year;

Exclusion Criteria:

1. Serious cardiac insufficiency, left ventricular ejection fraction<50;
2. Has a history of severe pulmonary function damaging;
3. Merging other malignant tumor;
4. Merging uncontrolled infection;
5. Merging the metabolic diseases (except diabetes);
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. patients with active hepatitis B or hepatitis C;
8. patients with HIV infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Happened in 3 ~ 4 acute GvHD after allogeneic hematopoietic stem cell transplantation on recurring patients;
11. Pregnancy or lactation women;
12. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety | 28 days
  Number of Participants with Severe/Adverse Events as a Measure of Safety
CAR-T Cell expansion level | 24 months
  Copies numbers of CAR in peripheral blood(PB) and/or bone marrow(BM)

SECONDARY OUTCOMES:
Objective response rate of complete remission and partial remission | 24 months
  Objective response rate of complete remission and partial remission
Overall survival time | 24 months
  Overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin luo, PhD&MD, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- No.2 Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No